CLINICAL TRIAL: NCT03334916
Title: A Randomized, Double-Blind, Placebo-Controlled, Multicenter Trial to Evaluate the Efficacy and Safety of YMC026 in Respiratory Disease Patients With Cough and Sputum as the Main Symptoms
Brief Title: A Clinical Trial to Evaluate the Efficacy and Safety of YMC026 in Respiratory Disease Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YMC026
Record Dates: First submitted 2017-10-31; First posted 2017-11-07 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Respiratory Disease
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- YMC026 (Experimental): 108 subjects will be assigned in this group. They will be administered 20mL of YMC026 three times a day for 6 days.
  Interventions: Drug: YMC026
- Placebo (Placebo Comparator): 108 subjects will be assigned in this group. They will be administered 20mL of placebo three times a day for 6 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: YMC026 — YMC026 20mL TID
  Arms: YMC026
Drug: Placebo — Placebo 20mL TID
  Arms: Placebo

SUMMARY:
This is a phase 4, randomized, double-blind, multicenter clinical trial to evaluate the efficacy and safety of YMC026 in respiratory disease patients with cough and sputum as the main symptoms

DETAILED DESCRIPTION:
The study has planned 4 visits during 2 weeks period (1 week of screening period, 1 week of treatment period). All subjects who agree to participate in the study and voluntarily give written informed consent are assessed by inclusion and exclusion criteria at the screening visit. After the screening period, the final eligibility of the subjects will be assessed at the randomization visit. Subjects who are determined to be appropriate for this study will be allocated to experimental group(YMC026) or control group(placebo) randomly in a 1:1 ratio. Subject will be administered the investigational product daily for 6 days. The safety for the subjects will be assessed at Day 3 and Day 6 visit, and the efficacy evaluation will be assessed at Day 6 visit.

ELIGIBILITY:
Inclusion Criteria:

1. Both gender, 15 years ≤ age < 75 years
2. Patients with BSS(Bronchitis Severity Score) ≥ 5point at screening visit and randomization visit
3. Written consent voluntarily to participate in this clinical trial

Exclusion Criteria:

1. Patients with severe respiratory disease
2. Patients with severe pulmonary disease
3. Patients who has history for drug hypersensitivity or allergic reaction in component of investigational product or similar drug
4. Patients with pregnant and/or have breast feeding
5. Patients who were treated with monoamine oxidase inhibitor, antihistamines, anti-viral drugs and glucocorticoids within 2 weeks prior to administration of investigational product
6. Patients who were treated with β2-agonist and anticholinergic drug within 1 weeks prior to administration of investigational product
7. Patients who were treated with secretolytics, mucolytics and bronchodilators within 1 day prior to administration of investigational product
8. Patients who are participating in another trial within 30 days prior to screening visit
9. Patients who investigators determines not appropriate to take part in this clinical study

Ages: 15 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 223 (Actual)
Dates: Start 2017-10-27 (Actual); Primary Completion 2018-04-11 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Change from Baseline BSS at Day 6 | Baseline(Day 0), Day 6
  Bronchitis Severity Score

SECONDARY OUTCOMES:
Change from Baseline BCSS at Day 6 | Baseline(Day 0), Day 6
  Breathlessness, Cough, and Sputum Scale
Patients´ evaluation of symptoms of cough and sputum on patient's diary | Day 6

CONTACTS AND LOCATIONS:
Locations (1):
- The Catholic University of Korea, Seoul St.Mary's Hospital, Seoul, South Korea